CLINICAL TRIAL: NCT04631315
Title: Efficacy and Safety of Difluprednate Ophthalmic Emulsion vs. a Fixed-Combination of Prednisolone Acetate - Phenylephrine Ophthalmic Suspension on Post-operative Inflammation Following Cataract Surgery.
Brief Title: Difluprednate vs. a Prednisolone Acetate - Phenylephrine on Post-operative Inflammation Following Cataract Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Poen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIFLUPRED03
Record Dates: First submitted 2020-11-05; First posted 2020-11-17 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2020-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — OmpF protein; prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Difluprednate Ophthalmic Emulsion 0.05%
  Interventions: Drug: Difluprednate Ophthalmic Emulsion 0.05%
- Comparator (Active Comparator): Prednisolone Acetate 1% - Phenylephrine 0.12% Ophthalmic Suspension
  Interventions: Drug: Prednisolone Acetate 1% Phenylephrine hydrochloride 0,12% ophthalmic solution

INTERVENTIONS:
Drug: Difluprednate Ophthalmic Emulsion 0.05% — 1 drop, 2 times a day, starting the day before surgery and continuing for 14 post-surgical days and 1 drop, once a day for the next 2 weeks.
  Other Names: Tolf®
  Arms: Intervention
Drug: Prednisolone Acetate 1% Phenylephrine hydrochloride 0,12% ophthalmic solution — 1 drop, 4 times a day, starting the day before surgery and continuing for 14 post-surgical days and 1 drop, twice a day for the next 2 weeks.
  Arms: Comparator

SUMMARY:
This controlled, randomized, double blind, multicenter study will be carried out to demonstrate that the topical ophthalmic nanoemulsion of difluprednate 0.05% (Tolf®, Poen Laboratories), has a high anti-inflammatory efficacy, which would allow it to be administered after cataract surgery 1 drop, twice a day , starting the day before surgery and continuing for 14 days and 1 drop, once a day for the following 2 weeks, achieving an adequate anti-inflammatory activity, with the benefit of reducing the toxicity on the ocular surface, improving the dosage and adherence to treatment.

The follow-up time will be 28 days and the outcome measures will be evaluated in a baseline (time 0), on day 1, on day 4 and on day 28 after surgery. The active control will be prednisolone acetate 1% + phenylephrine hydrochloride 0.12% topical ophthalmic suspension (Prednefrin® Forte, Allergan Argentina) given 1 drop, 4 times a days and 1 drop, twice a day for the next 2 weeks. Corneal thickness, central macula thickness, endothelial cell count, intraocular pressure, visual acuity, anterior chamber clearance and lacrimal film recovery will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes between 45 and 65 years old (women who are not fertile) who undergo cataract surgery N2 and N3, defined according to BCN10, Decimal classification of cataracts.
* That the surgical technique is ultrasonic phacoemulsification.
* Patients who have an initial corneal thickness between 500 and 570 µm inclusive.
* Patients with initial intraocular pressure between 12 and 18 mm Hg inclusive.
* Patients with an endothelial cell count greater than 1000 cells / mm2

Exclusion Criteria:

* Patients who use eye medication, except eye lubricant.
* Patients who before surgery have not been able to dilate their pupil more than 5 mm
* Patients who have been treated with corticosteroids or systemic anti-inflammatory drugs for 2 weeks prior to enrollment
* Patients who have received periocular corticosteroid injections in the study eye within the previous 4 weeks or used depot corticosteroids within 2 months prior to enrollment
* Patients who have received a topical ocular corticosteroid or non-steroidal anti-inflammatory drug (NSAID) within 24 hours prior to enrollment
* History of glaucoma or ocular hypertension in the study eye, history or presence of endogenous uveitis, or corneal abrasion or ulceration
* Patients with a diagnosis or suspicion of keratoconjunctival disease caused by viruses, bacteria, or fungi
* Patients which presents an allergy to the drug to be tested or to any similar drug such as other corticosteroids
* History of increased intraocular pressure due to the use of corticosteroids
* Patients with pathological macular features
* Diabetics
* Breastfeeding women
* Patients with rheumatoid arthritis.
* Patients treated with Amiodarone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2019-03-24 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline corneal thickness between treatments | Baseline to visit 3 (96 hours from surgery)
  Demonstrate that 0.05% difluprednate ophthalmic nanoemulsion administered 1 drop, 2 times a day, beginning the day before cataract surgery and continuing for the first 14 postoperative days and then 1 drop, once a day for the next 14 days, it does not present an anti-inflammatory efficacy lower than treatment with prednisolone acetate 1% + phenylephrine hydrochloride 0.12% ophthalmic suspension administered 1 drop, 4 times a day starting the day before surgery and continuing during the first 14 post-surgical days and 1 drop , 2 times a day for the next 14 days, for the treatment of postsurgical inflammation, in patients operated on for N2 and N3 cataracts.
  Difluprednate 0.05% ophthalmic nanoemulsion will not be clinically inferior than Prednisolone acetate 1% + 0.12% phenylephrine hydrochloride ophthalmic suspension, if the difference in corneal thickness obtained with OCT between the baseline day and the post-surgical day it does not differ beyond 17 µm between treatments.

SECONDARY OUTCOMES:
Retinal Thickness | Day before surgery (-1); Day 1 after surgery (1); Day 4 after surgery (4); 28 days post surgery (28)
  Retinal Thickness measured by Optical Coherence Tomography (mm)
Corneal endothelial cell count | Day before surgery (-1); Day after surgery (1); Day 4 after surgery (4); 28 days post surgery (28).
  Corneal endothelial cell count measured by specular microscope (cells/mm2)
Visual acuity | Day before surgery (-1); Day after surgery (1); Day 4 after surgery (4); 28 days post surgery (28).
  Visual acuity measured by visual acuity standardized chart (20/20)
Flare and cell on anterior chamber | Day before surgery (-1); Day after surgery (1); Day 4 after surgery (4); 28 days post surgery (28).
  Presence of flare and cells on anterior chamber using slit lamp (biomicroscopy)
Intraocular pressure | Day before surgery (-1); Day after surgery (1); Day 4 after surgery (4); 28 days post surgery (28).
  Intraocular pressure measured by Goldmann tonometer (mmHg)
Equal safety profile of both treatments | Day before surgery (-1); Day 1 after surgery (1); Day 4 after surgery (4); 28 days post surgery (28)
  Report of adverse events of both treatments under study
Corneal Thickness by pachymetry | Day before surgery (-1); Day after surgery (1); Day 4 after surgery (4); 28 days post surgery (28).
  Corneal Thickness (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Tosi, M.D., Study Director — Laboratorios Poen
Locations (1):
- Laboratorios Poen, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No